CLINICAL TRIAL: NCT05408403
Title: Comparison of the Effects of Transversalis Fascia Plane Block and Anterior QLB ( TFPB and Anterior QLB ) on Postoperative Analgesia in Cesarean Section Surgery
Brief Title: Comparison of the Effects of TFPB and Anterior QLB on Postoperative Analgesia in Cesarean Section Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, SEZGİN BİLGİN, Medical Doctor, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: TFPB-QLB3
Record Dates: First submitted 2022-06-01; First posted 2022-06-07 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Analgesia; Acute Pain; Chronic Pain
Keywords: Regional Anesthesia; Acute and chronical pain; Transversalis Fascia Plane Block; Quadratus Lumborum Blocks; Cesarean Section
MeSH Terms: conditions — Agnosia; Acute Pain; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Randomization of the study will be done by a doctor who will not participate in patient follow-up with closed envelopes using computer-generated randomization codes.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The anesthesia doctor who will perform the interfascial plane block (TFPB, anterior QLB) will be informed with a sealed envelope by an independent assistant outside the study, and the patient will not know which block is performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transversalis Fascia Plane Block (Active Comparator): Transversalis Fascia Plane Block (TFPB) will be performed the patients in Group A after the cesarean section surgery. Patient controlled analgesia device (PCA) is used for all the patients in the first 24 hours postoperatively
  Interventions: Other: Regional anesthesia TFPB
- Quadratus Lumborum Block (Active Comparator): Anterior Quadratus Lumborum Block ( Anterior QLB) will be performed the patients in Group B after the cesarean section surgery. Patient controlled analgesia device (PCA) is used for all the patients in the first 24 hours postoperatively
  Interventions: Other: Regional anesthesia QLB

INTERVENTIONS:
Other: Regional anesthesia TFPB — Transversalis Fascia Plane Block will be performed with 25 mL of 0.25% bupivacaine,after the end of cesarean surgery before extubation.
  Other Names: Transversalis Fascia Plane Block
  Arms: Transversalis Fascia Plane Block
Other: Regional anesthesia QLB — Anterior Quadratus Lumborum Block will be performed with 25 mL of 0.25% bupivacaine, after the end of cesarean surgery before extubation.
  Other Names: Anterior Quadratus Lumborum Block
  Arms: Quadratus Lumborum Block

SUMMARY:
This study evaluates the postoperative analgesic effects of transversalis fascia plane block and anterior quadratus lumborum block in patients having cesarean section under general anesthesia. General anesthesia will be performed to all patients for the surgery.

DETAILED DESCRIPTION:
In this study, patients are divided into two groups. After the general anesthesia is performed and cesarean section surgery is over; TFPB block will be performed to patients in Group A ; while anterior QLB block will be performed to patients in Group B. In addition, patient controlled analgesia (PCA) will be used in the first 24 hours postoperatively. Group A - Patients in group A will have TFPB block after the surgery. In addition, patient controlled analgesia (PCA) will be used in the first 24 hours postoperatively. Group B - Patients in group B will have anterior QLB block after the surgery. In addition, patient controlled analgesia (PCA) will be used in the first 24 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Being pregnant for at least 37 weeks
* Planning an elective cesarean operation
* Being between the ages of 18-45

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) 3-4 patients with comorbidities (Serious renal, cardiac, hepatic disease)
* Being operated with spinal anesthesia
* Obesity (> 100 kg, BMI> 35 kg / m2)
* Contraindication of regional anesthesia (coagulopathy, abnormal international normalized ratio (INR), thrombocytopenia, infection at the injection site)
* Hypersensitivity to local anesthetics or a history of allergy
* Patients with a history of opioid use longer than four weeks
* Patients with psychiatric disorders
* Patients with anatomic deformity
* Patients who do not want to participate

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women planned for elective cesarean operation
Enrollment: 49 (Actual)
Dates: Start 2022-06-18 (Actual); Primary Completion 2022-09-18 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
Opioid consumption in the first 24 hours after surgery | Postoperative Day 1
  Morphine consumption in the first 24 hours will be counted by IV patient controlled analgesia device (PCA). Patients will be able to request opioids via PCA device when the nrs score is above 4.

SECONDARY OUTCOMES:
Post-operative acute pain | Postoperative Day 1
  Pain status will be evaluated based on numeric rating scale (NRS) scores at rest and after movement. Pain status will be evaluated at 1, 3, 6, 9, 12, 18, 24. hours after surgery. Each NRS is scores 0-10. (0=no pain ; 10=worst pain imaginable)
The time of first opioid requirement | Postoperative Day 1
  The time of first opioid requirement will be recorded during the postoperative first 24 hours

OTHER OUTCOMES:
The incidences of post-operative nausea and vomiting (PONV) | Postoperative Day 1
  the presence of nausea and vomiting will be recorded for 24 hours after surgery
The incidence of side effects related to local anesthetics, opioid use and regional anesthesia technic | Postoperative Day 1
  respiratory depression, local anesthetic (LA) toxicity, hematoma and organ damage.

CONTACTS AND LOCATIONS:
Overall Officials: Sezgin Bilgin, Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayıs University Faculty of Medicine, Samsun, Turkey (Türkiye)